CLINICAL TRIAL: NCT03502785
Title: An Open-Label, Multi-Center Trial of INO-5401 + INO-9012 in Combination With Atezolizumab in Subjects With Locally Advanced Unresectable or Metastatic/Recurrent Urothelial Carcinoma
Brief Title: INO-5401 + INO-9012 in Combination With Atezolizumab in Locally Advanced Unresectable or Metastatic/Recurrent Urothelial Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCa-001
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — rocakinogene sifuplasmid; atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Cohort A (Experimental): Participants with locally advanced unresectable or metastatic/recurrent UCa, who have confirmed disease progression during or following treatment with an anti-PD-1/PD-L1 therapy. Cohort A participants will be treated with INO-5401 and INO-9012 in combination with atezolizumab.
  Interventions: Biological: INO-5401; Biological: INO-9012; Drug: Atezolizumab; Device: CELLECTRA™ 2000
- Cohort B (Experimental): Participants with locally advanced unresectable or metastatic/recurrent UCa who are treatment naïve and ineligible for cisplatin-based chemotherapy. Cohort B participants will be treated with INO-5401 and INO-9012 in combination with atezolizumab.
  Interventions: Biological: INO-5401; Biological: INO-9012; Drug: Atezolizumab; Device: CELLECTRA™ 2000

INTERVENTIONS:
Biological: INO-5401 — INO-5401 (9 milligram [mg] dose IM): mixture of 3 synthetic plasmids that target Wilms' tumor gene-1 (WT1) antigen, prostate-specific membrane antigen (PSMA) and human telomerase reverse transcriptase (hTERT) antigen.
Biological: INO-9012 — INO-9012 (1 mg dose IM): A synthetic plasmid that expresses human interleukin-12 (IL-12).
  INO-5401 + INO-9012 will be administered IM followed by EP with CELLECTRA™ 2000 device every 3 weeks for 4 doses then every 6 weeks for 6 additional doses, thereafter every 12 weeks until confirmed disease progression, unacceptable toxicity, or deemed intolerable by the investigator.
Drug: Atezolizumab — Atezolizumab will be administered by intravenous (IV) infusion every 3 weeks until confirmed disease progression, unacceptable toxicity, or deemed intolerable by the investigator.
Device: CELLECTRA™ 2000 — IM injection of INO-5401 and INO-9012 is followed by EP with the CELLECTRA™ 2000 device.

SUMMARY:
This is a Phase I/IIA, open-label, multi-center trial to evaluate the safety, immunogenicity and preliminary clinical efficacy of INO-5401 + INO-9012 delivered by intramuscular (IM) injection followed by electroporation (EP), in combination with atezolizumab in participants with locally advanced unresectable or metastatic/recurrent Urothelial Carcinoma (UCa). The trial population is divided into two cohorts: Cohort A: Participants with locally advanced unresectable or metastatic/recurrent UCa, who have confirmed disease progression during or following treatment with anti-Programmed Death receptor-1/Programmed Death receptor Ligand-1 (anti-PD-1/PD-L1) therapy; Cohort B: Participants with locally advanced unresectable or metastatic/recurrent UCa, who are treatment naïve and ineligible for cisplatin-based chemotherapy. A safety run-in will be performed with up to six participants (safety analysis participants) from cohort A.

ELIGIBILITY:
Inclusion Criteria:

* Sign an Informed Consent Form (ICF);
* Have histologically or cytologically documented locally advanced unresectable or metastatic/recurrent urothelial carcinoma (including renal pelvis, ureters, urinary bladder, and urethra);
* For Cohort A: Subjects who have radiographically confirmed disease progression during or following treatment with an anti-PD-1/PD-L1 based therapy;
* For Cohort B: No prior chemotherapy for inoperable locally advanced or metastatic or recurrent UCa and ineligible ("unfit") for cisplatin-based chemotherapy;
* Have measurable disease, as defined by RECIST version 1.1;
* Have a performance status of 0 or 1 on Eastern Cooperative Oncology Group (ECOG) Performance Scale;
* Have life expectancy of >/= 3 months;
* Be willing to provide a tissue sample for pre-treatment intra-tumoral assessment of proinflammatory and immunosuppressive factors;
* Have electrocardiogram (ECG) with no clinically significant findings as assessed by the investigator performed within 28 days prior to first dose;
* Demonstrate adequate hematological, renal, hepatic, and coagulation function;
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 5 months after the last dose of study treatment;
* For male subjects: agreement not to father a child. Participants must be surgically sterile (e.g, vasectomy) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 5 months after the last dose of study treatment.

Exclusion Criteria:

* Any approved anti-cancer therapy including chemotherapy, targeted small molecule therapy or radiation therapy within 2 weeks prior to trial Day 0 as well as current participation or recipient of treatment on a clinical trial within 28 days prior to Day 0;
* Documented active or untreated central nervous system (CNS) metastases and/or carcinomatous meningitis;
* Malignancies other than UCa within 3 years prior to Day 0, with the exception of those with negligible risk of metastasis or death treated with expected curative outcome;
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies;
* Treatment with systemic immunostimulatory agents;
* Treatment with systemic immunosuppressive medication;
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins;
* Known hypersensitivity allergy or contraindication to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the PD-1/PD-L1 inhibitor formulation;
* Active or history of autoimmune disease or immune deficiency;
* History or any evidence of interstitial lung disease;
* History of human immunodeficiency virus (HIV);
* Active hepatitis B or active hepatitis C;
* Severe infections within 4 weeks prior to enrollment;
* Received therapeutic oral or IV antibiotics within 2 weeks prior to Day 0;
* History or current evidence of any condition, therapy or laboratory abnormality that might confound the results of the trial; interfere with the subject's participation for the full duration of the trial, or is negatively impacted by EP treatment, or is not in the best interest of the subject to participate in the opinion of the treating investigator;
* Prior allogeneic stem cell or solid organ transplant;
* Uncontrolled tumor-related pain; pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures; or, hypercalcemia or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | From baseline up to 90 days after last dose of study medication (up to approximately 2 years and 3 months)
Antigen-Specific Cellular Immune Response | At baseline, Weeks 3, 6, 9, 12 and every 12 weeks thereafter up to end of study (up to approximately 2 years)
Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by Investigator Review in Cohort A | From Baseline to disease progression or death, whichever occurs first (up to approximately 2 years)

SECONDARY OUTCOMES:
ORR by RECIST version 1.1 by Investigator Review in Cohort B | From Baseline to disease progression or death, whichever occurs first (up to approximately 2 years)
ORR by Immune RECIST (iRECIST) | From Baseline to disease progression or death, whichever occurs first (up to approximately 2 years)
Duration of Response (DoR) | From Baseline to disease progression or death, whichever occurs first (up to approximately 2 years)
Progression Free Survival (PFS) as Assessed by RECIST version 1.1 and iRECIST | From Baseline to disease progression or death, whichever occurs first (up to approximately 2 years)
Overall Survival (OS) | : From Baseline to the time of death from any cause (up to approximately 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Skolnik, MD, Study Director — Inovio Pharmaceuticals
Locations (11):
- United States (11):
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - H. Lee Moffitt Cancer Center & Research Institute, Inc., Tampa, Florida
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - New York University Langone Medical Center - Perlmutter Cancer Center, New York, New York
  - Columbia University, Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Inova Melanoma and Skin Cancer Center, Fairfax, Virginia